CLINICAL TRIAL: NCT02514382
Title: A Phase 1b Study of REOLYSIN® (Reovirus Serotype 3 - Dearing Strain) Combined With Standard Doses of Bortezomib and Dexamethasone in Patients With Relapsed/Refractory Multiple Myeloma
Brief Title: Wild-Type Reovirus, Bortezomib, and Dexamethasone in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Oncolytics Biotech (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16M-15-2; NCI-2015-01069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); REO 019; 16M-15-2 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-07-30; First posted 2015-08-03 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Recurrent Plasma Cell Myeloma; Refractory Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; reolysin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (dexamethasone, bortezomib, wild-type reovirus) (Experimental): Patients receive dexamethasone PO, IV, or IM and bortezomib SC (preferably) or IV over 3-5 seconds on days 1, 8, and 15. Patients also receive wild-type reovirus IV over 60 minutes on days 1, 2, 8, 9, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Biological: Wild-type Reovirus

INTERVENTIONS:
Drug: Bortezomib — Given SC or IV
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Drug: Dexamethasone — Given PO, IV, or IM
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Biological: Wild-type Reovirus — Given IV
  Other Names: Reolysin

SUMMARY:
This phase Ib trial studies the safety and best dose of wild-type reovirus in combination with bortezomib and dexamethasone and to see how well they work in treating patients with multiple myeloma that has returned (relapsed) or does not respond to treatment (refractory). A virus, called wild-type reovirus, may be able to infect cancer cells and slow the cancer growth and kill cancer cells. Bortezomib and dexamethasone may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving wild-type reovirus together with bortezomib and dexamethasone may be a better treatment for multiple myeloma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) with the maximum REOLYSIN (wild-type reovirus) dose limited to 4.5 x 10^10 tissue culture infection dose (TCID)50 and the safety profile of REOLYSIN in combination with bortezomib and dexamethasone in patients with relapsed or refractory multiple myeloma (MM). (Phase 1b) II. To further explore the safety and tolerability of the combination and to determine the overall response rate (ORR) (complete response [CR] + partial response [PR]) to REOLYSIN in combination with bortezomib and dexamethasone in patients with relapsed or refractory MM. (Phase 1b Dose Expansion)

SECONDARY OBJECTIVES:

I. To determine ORR in the Phase 1b part to the combination at escalating doses.

II. To determine the progression-free survival (PFS) of patients with relapsed or refractory MM treated with REOLYSIN in combination with bortezomib and dexamethasone.

III. To evaluate the effect of REOLYSIN in combination with bortezomib and dexamethasone treatments on overall survival (OS).

IV. To conduct pharmacodynamic studies as described.

OUTLINE: This is a phase Ib, dose-escalation study of wild-type reovirus followed by a phase Ib expansion trial.

Patients receive dexamethasone orally (PO), intravenously (IV), or intramuscularly (IM) and bortezomib subcutaneously (SC) (preferably) or IV over 3-5 seconds on days 1, 8, and 15. Patients also receive wild-type reovirus IV over 60 minutes on days 1, 2, 8, 9, 15, and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 1 month and then every 3 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Have relapsed or refractory MM after at least one line of therapy
* Have a confirmed diagnosis of MM with measurable disease, as defined by the presence of monoclonal immunoglobulin protein in serum electrophoreses of at least 0.5 g/dL for immunoglobulin G (IgG) or 0.25 g/dL for IgA, or measurable light chain in serum (100 mg/L) or urinary excretion of at least 200 mg monoclonal light chain per 24 hours
* Have NO continuing acute toxic effects (except alopecia) of any prior chemotherapy, radiotherapy or surgical procedures; all such effects must have resolved to Common Terminology Criteria for Adverse Events (CTCAE, Version 4.03) grade =< 1; surgery (except minor procedures such as biopsies, IV line placement, etc.) must have occurred at least 28 days prior to study enrollment
* Have received NO anti-cancer therapy within 28 days prior to receiving study drug
* Have received NO radiotherapy within 14 days prior to receiving study drug
* Have an Eastern Cooperative Oncology Group (ECOG) Performance score =< 2
* Have a life expectancy of at least 3 months
* Absolute neutrophil count (ANC) >= 1 x 10^9 (International System [SI] units 10^9/L) (with or without filgrastim [G-CSF])
* Platelets >= 50 x10^9 (SI units 10^9/L)
* Serum creatinine =< 2 x upper limit of normal (ULN)
* Bilirubin =< 1.5 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 3 x ULN (=< 5 x ULN if patients have liver involvement with MM)
* Proteinuria < grade 2
* Have a negative pregnancy test if a female with childbearing potential
* Have signed an informed consent indicating that the patient is aware of the neoplastic nature of their disease and have been informed of the procedures of the protocol, the experimental nature of the therapy, possible alternative therapies, potential benefits, side effects, risks, and discomforts
* Be willing and able to comply with scheduled visits, the treatment plan, and laboratory tests

Exclusion Criteria:

* Have a history of or current evidence of intracranial disease; patients with brain metastases must be excluded from this clinical trial
* Be on immunosuppressive therapy or have human immunodeficiency virus (HIV) infection or active hepatitis B or C
* Be a pregnant or breast-feeding woman; female patients of childbearing potential must agree to use effective contraception, must be surgically sterile, or must be postmenopausal; male patients must agree to use effective contraception or be surgically sterile; barrier methods are a recommended form of contraception
* Have clinically significant cardiac disease (New York Heart Association, class III or IV) including pre-existing arrhythmia, uncontrolled angina pectoris, myocardial infarction 1 year prior to study entry, or a known history of grade 2 or higher compromised left ventricular ejection fraction
* Have dementia or altered mental status that would prohibit informed consent
* Have any other severe, acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the principal investigator, would make the patient inappropriate for this study
* Have a history of allergic (anaphylactic) sensitivity to bortezomib, boron or mannitol
* Have grade 2 or greater neuropathy at the time of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-08-21 (Actual); Primary Completion 2022-04-19 (Actual); Study Completion 2022-04-19 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events assessed by CTCAE version 4.03 | Up to 30 days post-treatment
  The safety of the bortezomib, dexamethasone, and wild-type reovirus combination will be assessed by the evaluation of the type, frequency, and severity of adverse events.

SECONDARY OUTCOMES:
ORR | Up to 3 years
  Will determine ORR (CR + PR) in the Phase 1b part to the combination at escalating doses.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Kelly, MD, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Nawrocki ST, Olea J, Villa Celi C, Dadrastoussi H, Wu K, Tsao-Wei D, Colombo A, Coffey M, Fernandez Hernandez E, Chen X, Nuovo GJ, Carew JS, Mohrbacher AF, Fields P, Kuhn P, Siddiqi I, Merchant A, Kelly KR. Comprehensive Single-Cell Immune Profiling Defines the Patient Multiple Myeloma Microenvironment Following Oncolytic Virus Therapy in a Phase Ib Trial. Clin Cancer Res. 2023 Dec 15;29(24):5087-5103. doi: 10.1158/1078-0432.CCR-23-0229. PMID 37812476